CLINICAL TRIAL: NCT01713868
Title: Social Media And Risk-reduction Training for Infant Care Practices (SMART)
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Yale University (Other); Boston University (Other)
Responsible Party: Principal Investigator, Rachel Moon, MD, Rachel Moon, M.D., University of Virginia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD072815-01 (NIH)
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Risk Reduction
Keywords: Breastfeeding; Safe Sleep; Messaging; Social Media
MeSH Terms: conditions — Risk Reduction Behavior; Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Safe Sleep Edu and Breastfeeding mHealth (Other): Participants will receive Safe Sleep Nursery Education and Breastfeeding Mobile Health messaging
  Interventions: Behavioral: Safe Sleep Nursery Education; Behavioral: Breastfeeding Mobile Health Messaging
- Breastfeeding Edu and Safe Sleep mHealth (Other): Participants will receive the Breastfeeding Nursery Education and the Safe Sleep Mobile Health messaging
  Interventions: Behavioral: Breastfeeding Nursery Education; Behavioral: Safe Sleep Mobile Health Messaging
- Safe Sleep Edu and Safe Sleep mHealth (Other): Participants will receive Safe Sleep Nursery Education and Safe Sleep Mobile Health messaging
  Interventions: Behavioral: Safe Sleep Nursery Education; Behavioral: Safe Sleep Mobile Health Messaging
- Breastfeed Edu and Breastfeed mHealth (Other): Participants will receive Breastfeeding Nursery Education and Breastfeeding Mobile Health messaging
  Interventions: Behavioral: Breastfeeding Nursery Education; Behavioral: Breastfeeding Mobile Health Messaging

INTERVENTIONS:
Behavioral: Safe Sleep Nursery Education — Nursery-based program for safe sleep
  Arms: Safe Sleep Edu and Breastfeeding mHealth; Safe Sleep Edu and Safe Sleep mHealth
Behavioral: Breastfeeding Nursery Education — Nursery-based program to promote breastfeeding
  Arms: Breastfeed Edu and Breastfeed mHealth; Breastfeeding Edu and Safe Sleep mHealth
Behavioral: Breastfeeding Mobile Health Messaging — Mobile messaging to provide multiple short culturally competent videos to promote breastfeeding delivered via email.
  Arms: Breastfeed Edu and Breastfeed mHealth; Safe Sleep Edu and Breastfeeding mHealth
Behavioral: Safe Sleep Mobile Health Messaging — Mobile messaging to provide multiple short culturally competent videos to promote safe sleep practices delivered via email.
  Arms: Breastfeeding Edu and Safe Sleep mHealth; Safe Sleep Edu and Safe Sleep mHealth

SUMMARY:
The goal of this proposal is to address serious and ongoing challenges related to adherence to public health recommendations known to reduce the risk of SIDS. Adherence has reached a plateau at an unacceptably low level both in the overall US population and especially in Black infants leading to a halt in the decline in infant mortality and a widening in the racial disparity in infant mortality. The current proposal is a collaborative effort that will capitalize on the extensive experience of the investigators in studying barriers to adherence to safe sleep practices to develop two complementary, culturally competent, intervention strategies and to test the effectiveness of each strategy as well as both strategies in combination. Innovative aspects of the Social Media and Risk-reduction Training of Infant Care Practices (SMART) study include its: 1) unique collaboration of leaders in the field; 2) leveraging of the currently operational infant care practices study infrastructure and hospitals; 3) use of two complementary interventions with the potential for synergistic impact; 4) use of social marketing strategies;5) use of mobile technology (mHealth) to deliver messages; and 6) collaboration with community resources and expertise. The SMART study will have four arms in which 16 hospitals are randomly assigned to one of the following study groups: 1) Safe Sleep Nursery Education and Breastfeeding mHealth messaging; 2) Breastfeeding Nursery Education and Safe Sleep mHealth messaging; 3) Safe Sleep Nursery Education and Safe Sleep mHealth messaging; 4) Breastfeeding Nursery Education and Breastfeeding mHealth messaging. A total of 1600 mothers will be recruited (100/hospital), with 400 in each study group. The primary aim is to assess the effectiveness of the interventions aimed at promoting safe sleep practices compared with the breastfeeding control interventions. The secondary aim is to assess potential mediating factors that may explain the intervention effects on infant care practices and that may inform areas for future improved intervention approaches. With the successful completion of the SMART study, effectiveness data will have been provided for two interventions to improve adherence to safe sleep practices that are practical to disseminate nationally in multiple diverse settings.

DETAILED DESCRIPTION:
FOA PAR-11-242 seeks research that will improve the design, implementation, and effectiveness of interventions to prevent Sudden Infant Death Syndrome (SIDS) and unintentional injury-related infant deaths associated with the sleep environment. The SMART (Social Media and Risk Reduction Training) Infant Care Practices proposal is a collaborative effort among researchers who collectively have generated much of the data on infant care practices that underlie the need for this FOA, and who have access to an already existing and operational infrastructure that permits performance of a large randomized clinical trial to study preventative interventions. This infrastructure was created for the NICHD-funded SAFE Infant Care Practices study, for which mothers are being recruited in 2011, 2012, and 2013 at a nationally-representative group of birth hospitals, with completion of infant care practice surveys at 2-5 months after birth. These hospitals, which will complete their participation in SAFE during 2013, are geographically and culturally diverse, will have had 3 years of baseline infant care practice data collected, and have a proven track record of successful recruitment. We will use our collective extensive experience studying barriers to adherence to safe sleep practices to develop two complementary, culturally competent intervention strategies and to test the effectiveness of each strategy, as well as both strategies in combination. Both of the proposed intervention strategies, described below, were selected largely because they can be used in diverse populations and offer the potential to be rapidly disseminated nationwide.

Nursery Education: A nursery-based training program will be modeled after our successful pilot study and informed by our collective research on barriers to adopting safe sleep practices. We will use social marketing strategies to capture the attention of nursing staff and empower them to improve safe sleep practice modeling and messaging received by mothers and extended families during the post-partum hospital stay.

mHealth: We will use an innovative approach, using mobile messaging, that applies expertise in social marketing to provide multiple short culturally competent videos delivered via email from the end of the post-partum hospital stay through 2 months of age. This strategy will leverage the internet as a powerful tool to access health information, and mobile devices (e.g., cell phones), which have made internet access possible for many, particularly those who are younger, minority, and from lower socioeconomic and educational backgrounds. Using technology to deliver health-related information is likely to be a well-accepted and effective strategy, particularly among minority and low-income populations. Indeed, studies demonstrate that email may be an effective, inexpensive, and time-efficient strategy to transmit health information.

For each of the safe sleep practice interventions (Nursery Education and mHealth), we will develop control interventions in which the Nursery Education or mHealth approach is used to promote breastfeeding. We have chosen breastfeeding as the control intervention because it 1) is not expected to impact endpoints critical to the assessment of the safe sleep practice intervention, and 2) provides health promoting messages to control mothers.

In the SMART study, we propose a 4-arm RCT in which 16 hospitals completing participation in the SAFE study are randomly assigned to one of the following groups (with Safe Sleep Intervention and/or Breastfeeding Control): 1) Safe Sleep Nursery Education and Breastfeeding mHealth messaging; 2) Breastfeeding Nursery Education and Safe Sleep mHealth messaging; 3) Safe Sleep Nursery Education and Safe Sleep mHealth messaging; and 4) Breastfeeding Nursery Education and Breastfeeding mHealth messaging. We are uniquely positioned to design, implement and test the effectiveness of these interventions in a methodologically rigorous way and propose the following specific aims: Primary Aim: To assess the effectiveness of the interventions aimed at promoting safe sleep practices compared with the breastfeeding controls.

Hypothesis:For each recommended safe sleep practice (supine sleep position, not bed sharing, pacifier use, avoiding use of soft bedding), when controlling for other variables, there will be: a) an increased adherence for mothers who received Safe Sleep Nursery Education; b) an increased adherence for mothers who received Safe Sleep mHealth messaging; and c) compared to mothers who received either Safe Sleep Nursery Education or Safe Sleep mHealth messaging alone, an increased adherence for mothers who received both Safe Sleep Nursery Education and Safe Sleep mHealth messaging.

Secondary Aim: Assess potential mediating factors that may explain the intervention effects on infant care practices and that may inform areas for future improved intervention approaches.

Hypothesis: Changes in variables within each of the domains of the Theory of Planned Behavior (Attitudes/Beliefs, Social Norms, Perceived Control) will be mediators of the effectiveness of safe sleep interventions.

ELIGIBILITY:
Inclusion Criteria:

- mothers must live in the US, deliver a healthy infant in one of the study hospitals, plan to take her baby home with her, and be able to receive emails.

Exclusion Criteria:

- mothers who are not English speaking, whose infant is deceased, those not having custody of the infant, and those whose infants require hospitalization for more than 1 week, or have an ongoing medical problem requiring subspecialty care and mothers who are unable to receive email messages.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Corwin, MD, Principal Investigator — Boston University; Eve R Colson, M.D., Principal Investigator — Yale University; Fern R Hauck, M.D., M.S., Principal Investigator — University of Virginia; Rachel Moon, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kellams A, Kerr SM, Moon RY, Hauck FR, Heeren T, Colson E, Parker MG, Rice F, Corwin MJ. The Impact of Breastfeeding and Safe Sleep Mobile Health Messaging on Breastfeeding and Bedsharing. Acad Pediatr. 2022 Aug;22(6):927-934. doi: 10.1016/j.acap.2022.01.016. Epub 2022 Feb 4. PMID 35124281
- [Derived] Moon RY, Corwin MJ, Kerr S, Heeren T, Colson E, Kellams A, Geller NL, Drake E, Tanabe K, Hauck FR. Mediators of Improved Adherence to Infant Safe Sleep Using a Mobile Health Intervention. Pediatrics. 2019 May;143(5):e20182799. doi: 10.1542/peds.2018-2799. PMID 31015374
- [Derived] Moon RY, Hauck FR, Colson ER, Kellams AL, Geller NL, Heeren T, Kerr SM, Drake EE, Tanabe K, McClain M, Corwin MJ. The Effect of Nursing Quality Improvement and Mobile Health Interventions on Infant Sleep Practices: A Randomized Clinical Trial. JAMA. 2017 Jul 25;318(4):351-359. doi: 10.1001/jama.2017.8982. PMID 28742913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
Started | 400 | 400 | 400 | 400
Completed | 303 | 335 | 320 | 305
Not Completed | 97 | 65 | 80 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth | Total
Number analyzed (Participants) | 400 | 400 | 400 | 400 | 1600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 14 | 42 | 21 | 109
  Between 18 and 65 years | 368 | 386 | 358 | 379 | 1491
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (5.9) | 29.3 (5.8) | 27.1 (5.9) | 27.6 (5.7) | 27.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number of participants with data to analyze differed from the number of participants recruited because of attrition.
  Participants
    number analyzed (Participants) | 303 | 335 | 320 | 305 | 1263
    Female | 303 | 335 | 320 | 305 | 1263
    Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 128 | 121 | 144 | 127 | 520
  Not Hispanic or Latino | 272 | 279 | 256 | 273 | 1080
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 26 | 6 | 20 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 173 | 101 | 95 | 133 | 502
  White | 112 | 205 | 187 | 141 | 645
  More than one race | 20 | 11 | 7 | 8 | 46
  Unknown or Not Reported | 83 | 57 | 105 | 98 | 343
Maternal educational level [Count of Participants; unit: Participants] — Population: Because of attrition, number analyzed is less than number recruited.
  Participants
    number analyzed (Participants) | 303 | 335 | 320 | 305 | 1263
    Less than high school | 36 | 11 | 31 | 10 | 88
    High school or GED | 84 | 63 | 77 | 88 | 312
    Some college | 102 | 114 | 118 | 104 | 438
    College or more | 80 | 147 | 92 | 101 | 420
    Unknown | 1 | 0 | 2 | 2 | 5
Household income [Count of Participants; unit: Participants] — Population: Because of attrition, number analyzed is less than number recruited
  Participants
    number analyzed (Participants) | 303 | 335 | 320 | 305 | 1263
    Less than $20,000 | 49 | 30 | 55 | 47 | 181
    $20,000-49.999 | 59 | 62 | 56 | 62 | 239
    $50,000 or more | 81 | 175 | 91 | 88 | 435
    Unknown | 114 | 68 | 118 | 108 | 408
Maternal marital status [Count of Participants; unit: Participants] — Population: Because of attrition, number analyzed is less than number recruited
  Participants
    number analyzed (Participants) | 303 | 335 | 320 | 305 | 1263
    Married | 127 | 203 | 147 | 163 | 640
    Never married | 158 | 111 | 151 | 132 | 552
    Divorced, separated, or widowed | 14 | 20 | 14 | 8 | 56
    Unknown | 4 | 1 | 8 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Recommended Supine Sleep Position
Description: Hypothesis:For supine sleep position, when controlling for other variables, there will be: a) an increased adherence for mothers who received Safe Sleep Nursery Education; b) an increased adherence for mothers who received Safe Sleep mHealth messaging; and c) compared to mothers who received either Safe Sleep Nursery Education or Safe Sleep mHealth messaging alone, an increased adherence for mothers who received both Safe Sleep Nursery Education and Safe Sleep mHealth messaging. Outcome measures will be assessed by survey conducted when the infant is 2-5 months of age.
Time Frame: 6 months
Population: Results analyzed at 2+ months infant age.
Measure: Count of Participants; unit: Participants
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
Number analyzed (Participants) | 301 | 333 | 319 | 303
Participants
  Usual supine sleep position | 230 | 294 | 294 | 243
  Usual nonsupine position | 71 | 39 | 25 | 60
Statistical Analysis 1: Comparison: Safe Sleep Edu and Breastfeeding mHealth vs Breastfeeding Edu and Safe Sleep mHealth vs Safe Sleep Edu and Safe Sleep mHealth vs Breastfeed Edu and Breastfeed mHealth; Sample size provided power of detecting the effect of an individual intervention in the presence of interaction.We assumed pre-study prevalence of a safe sleep practice ranging from 50% to 60% across hospitals. We powered the study to detect a 10 percentage point difference between two study groups, and determined that an analysis sample of n=1280 (320 per treatment group) was needed for 80% power (testing at two-sided p<0.05). Allowing for 20% loss to follow-up, this led to a sample of n=1600; Test type: Superiority — GEE logistic regression accounted for within-hospital clustering, individual-level & hospital-level covariates. We converted aORs to aRDs (95% CI) using the BF/BF group as the control group prevalence and reported separate effects of the 2 interventions. We fit multiplicative interaction models with indicator variables for education, mHealth, and their interaction. As the interaction between interventions was significant, we presented results from the interaction model; p = 0.03, Regression, Logistic — Adjusted education effect p=0.34. Adjusted mHealth effect p<0.001. Test for interaction p=0.01. Adjusted education only effect p=0.74. Adjusted mHealth only effect p=0.02. Adjusted mHealth and education effect: p=0.03

2. Primary Outcome: Adherence With Recommended Roomsharing Without Bed Sharing
Description: Hypothesis: For roomsharing without bed sharing, when controlling for other variables, there will be: a) an increased adherence for mothers who received Safe Sleep Nursery Education; b) an increased adherence for mothers who received Safe Sleep mHealth messaging; and c) compared to mothers who received either Safe Sleep Nursery Education or Safe Sleep mHealth messaging alone, an increased adherence for mothers who received both Safe Sleep Nursery Education and Safe Sleep mHealth messaging. Outcome measures will be assessed by survey conducted when the infant is 2-5 months of age.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
Number analyzed (Participants) | 293 | 328 | 313 | 291
Participants
  Roomsharing without bedsharing | 218 | 262 | 269 | 205
  Not roomsharing without bedsharing | 75 | 66 | 44 | 86
Statistical Analysis 1: Comparison: Safe Sleep Edu and Breastfeeding mHealth vs Breastfeeding Edu and Safe Sleep mHealth vs Safe Sleep Edu and Safe Sleep mHealth vs Breastfeed Edu and Breastfeed mHealth; Sample size provided power of detecting the effect of an individual intervention in the presence of interaction. We assumed pre-study prevalence of a safe sleep practice ranging from 50% to 60% across hospitals. We powered the study to detect a 10 percentage point difference between two study groups, and determined that an analysis sample of n=1280 (320 per treatment group) was needed for 80% power (testing at two-sided p<0.05). Allowing for 20% loss to follow-up,this led to a sample of n=1600; Test type: Superiority — GEE logistic regression accounted for within-hospital clustering, individual-level & hospital-level covariates. We converted aORs to aRDs (95% CI) using the BF/BF group as the control group prevalence and reported separate effects of the 2 interventions. We fit multiplicative interaction models with indicator variables for education, mHealth, and their interaction. As the interaction between interventions was not significant, we only presented main effects model; p < 0.001, Regression, Logistic — Adjusted education effect: p=0.22. Adjusted mHealth effect p<0.001. Test for interaction p=0.08

3. Primary Outcome: Adherence With Recommended Pacifier Use
Description: Hypothesis: For pacifier use, when controlling for other variables, there will be: a) an increased adherence for mothers who received Safe Sleep Nursery Education; b) an increased adherence for mothers who received Safe Sleep mHealth messaging; and c) compared to mothers who received either Safe Sleep Nursery Education or Safe Sleep mHealth messaging alone, an increased adherence for mothers who received both Safe Sleep Nursery Education and Safe Sleep mHealth messaging. Outcome measures will be assessed by survey conducted when the infant is 2-5 months of age.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
Number analyzed (Participants) | 290 | 326 | 315 | 291
Participants
  Usual pacifier use | 193 | 226 | 240 | 174
  Usual no pacifier use | 97 | 100 | 75 | 117
Statistical Analysis 1: Comparison: Safe Sleep Edu and Breastfeeding mHealth vs Breastfeeding Edu and Safe Sleep mHealth vs Safe Sleep Edu and Safe Sleep mHealth vs Breastfeed Edu and Breastfeed mHealth; Sample size provided power of detecting the effect of an individual intervention in the presence of interaction. We assumed pre-study prevalence of a safe sleep practice ranging from 50% to 60% across hospitals. We powered the study to detect a 10 percentage point difference between two study groups, and determined that an analysis sample of n=1280 (320 per treatment group) was needed for 80% power (testing at two-sided p<0.05). Allowing for 20% loss to follow-up, this led to a sample of n=1600; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Logistic — Adjusted education effect p=0.07. Adjusted mHealth effect p<0.001. Test for interaction p=0.54

4. Primary Outcome: Adherence With Recommended Avoiding Use of Soft Bedding
Description: Hypothesis: For each recommended avoidance of soft bedding use, when controlling for other variables, there will be: a) an increased adherence for mothers who received Safe Sleep Nursery Education; b) an increased adherence for mothers who received Safe Sleep mHealth messaging; and c) compared to mothers who received either Safe Sleep Nursery Education or Safe Sleep mHealth messaging alone, an increased adherence for mothers who received both Safe Sleep Nursery Education and Safe Sleep mHealth messaging. Outcome measures will be assessed by survey conducted when the infant is 2-5 months of age.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
Number analyzed (Participants) | 300 | 333 | 320 | 299
Participants
  No soft bedding use | 204 | 259 | 262 | 202
  Soft bedding use | 96 | 74 | 58 | 97
Statistical Analysis 1: Comparison: Safe Sleep Edu and Breastfeeding mHealth vs Breastfeeding Edu and Safe Sleep mHealth vs Safe Sleep Edu and Safe Sleep mHealth vs Breastfeed Edu and Breastfeed mHealth; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Regression, Logistic — Adjusted education effect p=0.33. Adjusted mHealth effect p<0.001. Test for interaction p=0.29

5. Secondary Outcome: Number of Participants Reporting Positive/Nonpositive Attitudes Towards Supine Sleep
Description: Questions assessing attitudes toward sleep position included the mothers' ratings regarding if she believed that each infant sleep position (back, side, stomach) made the baby healthy, safer, more comfortable, and kept the baby from choking. Positive attitudes were defined as having positive attitudes toward the recommended behavior AND not having positive attitudes toward other behaviors (e.g., having positive attitudes towards both supine and side sleep would lead to a categorization of not having positive attitudes towards supine sleep only).
Time Frame: 6 months
Population: All 4 arms received a combination of education (breastfeeding or safe sleep) and mHealth (breastfeeding or safe sleep). Only the mHealth interventions were effective. Thus, for this analysis, we collapsed the arms to 2 arms: received mHealth breastfeeding and received mHealth safe sleep.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Received mHealth breastfeeding
- mHealth Safe Sleep: Received mHealth safe sleep
Arm/Group | Control | mHealth Safe Sleep
Number analyzed (Participants) | 608 | 655
Participants
  # reporting positive attitudes re supine sleep | 313 | 491
  # reporting nonpositive attitudes re supine sleep | 295 | 164
Statistical Analysis 1: Comparison: Control vs mHealth Safe Sleep; Test type: Other — Causal mediation analysis; Difference in proportions = 0.16; We performed causal mediation analyses to estimate the Total Effect of intervention on a categorical outcome as the difference in the proportion with the outcome for those who received the intervention and were positive on the mediator vs. those who received the control and were negative on the mediator. Significance is determined through 95% confidence intervals (CIs), with CIs not including 0.0 indicating significant effects

6. Secondary Outcome: Number of Participants Reporting Positive/Nonpositive Attitudes Towards Roomsharing Without Bedsharing.
Description: Questions assessing attitudes toward sleep location (bedsharing, roomsharing without bedsharing) assessed whether the location was pleasant for the baby and/or mother, safer for the baby, more comfortable for the baby and/or mother, and kept the baby from choking. Positive attitudes were defined as having positive attitudes toward the recommended behavior AND not having positive attitudes toward other behaviors (e.g., having positive attitudes towards both bedsharing and not bedsharing would lead to a categorization of not having positive attitudes towards bedsharing only).
Time Frame: 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Control | mHealth Safe Sleep
Number analyzed (Participants) | 608 | 655
Participants
  Positive attitude re: roomsharing w/o bedsharing | 306 | 442
  Nonpositive attitude re roomsharing w/o bedsharing | 302 | 213
Statistical Analysis 1: Comparison: Control vs mHealth Safe Sleep; Test type: Other — Causal mediation analysis; Difference in proportions = 0.14; [other analysis details as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants Reporting Positive/Nonpositive Social Norms re Supine Sleep
Description: Social norms were assessed by asking if the people most important to the mother thought that the baby should sleep in each position or location. Positive social norms were defined as having positive norms toward the recommended behavior AND not having positive norms toward other behaviors.
Time Frame: 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Control | mHealth Safe Sleep
Number analyzed (Participants) | 608 | 655
Participants
  Positive social norms re supine sleep | 332 | 466
  Nonpositive social norms re supine sleep | 276 | 189
Statistical Analysis 1: Comparison: Control vs mHealth Safe Sleep; Test type: Other — Causal mediation analysis; Difference in proportions = 0.14; [other analysis details as in outcome 5, analysis 1]

8. Secondary Outcome: Number of Participants Reporting Positive/Nonpositive Social Norms re: Roomsharing Without Bedsharing.
Description: as for outcome 7
Time Frame: 6 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Control | mHealth Safe Sleep
Number analyzed (Participants) | 608 | 655
Participants
  Positive social norms re roomsharing w/o bedsharin | 297 | 350
  Nonpositive norms re roomsharing w/o bedsharing | 311 | 305
Statistical Analysis 1: Comparison: Control vs mHealth Safe Sleep; Test type: Other — Causal mediation analysis; Difference in proportions = 0.15; [other analysis details as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Safe Sleep Edu and Breastfeeding mHealth | Breastfeeding Edu and Safe Sleep mHealth | Safe Sleep Edu and Safe Sleep mHealth | Breastfeed Edu and Breastfeed mHealth
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/400 | 0/400 | 0/400
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/400 | 0/400
Other Adverse Events (participants affected / at risk) | 0/400 | 0/400 | 0/400 | 0/400

LIMITATIONS AND CAVEATS:
There was a 21% loss to follow-up, not generalizable to non-English-speaking populations, not powered to assess adverse events, did not measure clinical outcomes (i.e., rates of sudden unexpected infant death), and the results were self-reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No